CLINICAL TRIAL: NCT05839223
Title: Clinical Pharmacist Role in Increasing the Adherence to Recommendations Among Patients Using Isotretinoin: A Randomized, Controlled Study
Brief Title: Clinical Pharmacist Role in Adherence to Recommendations Among Isotretinoin Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bushra Mahmoud Ahmad Hijazi, Assistant Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IsoJordanUST
Record Dates: First submitted 2023-03-12; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Acne Vulgaris
Keywords: Isotretinoin, Clinical Pharmacist, Counseling, Adherence
MeSH Terms: conditions — Acne Vulgaris | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): received the educational process (recommendations) about isotretinoin by a clinical pharmacist in addition to the routine education about isotretinoin provided by the physician
  Interventions: Other: Education
- Control (No Intervention): received only the routine education about isotretinoin provided by the physician

INTERVENTIONS:
Other: Education — educational process (recommendations) about isotretinoin by a clinical pharmacist.
  The information included: the degree of the importance of adherence to the drug and the recommendations, the correct method of taking it, the importance of doing periodic laboratory tests (lipid profile, liver enzyme test, and pregnancy test), common side effects, how to properly avoid and deal with side effects, precaution warnings they should pay attention to, and what are the cases in which the drug should be stopped.
  Arms: Intervention

SUMMARY:
The objective of the study was to evaluate the role of clinical pharmacists in improving adherence to medication and the recommendations related to isotretinoin, awareness about proper use, dealing with the side effects, and anxiety and depressive symptoms. Patients were randomly assigned to an intervention group (received the educational process (recommendations) about isotretinoin by a clinical pharmacist in addition to the routine education about isotretinoin provided by the physician) and a control group (received only the routine education about isotretinoin provided by the physician) and then followed for three months. Patient's adherence to the recommendations, patient's knowledge about isotretinoin, and side effects management for both groups were measured through a set of questions adapted from a validated questionnaire at baseline and after three months. Adherence scale was used to evaluate adherence to the medication after three months. Hospital Anxiety and Depression Scale were used to assess depressive and anxiety symptoms at baseline and at follow-up in each group.

DETAILED DESCRIPTION:
Patients and Settings

Patients who attended dermatological clinics (at King Abdullah University Hospital (KAUH), Princess Basma Hospital (PBH), and Prince Rashid Hospital (PRH). The study was conducted over the period from September/2020 to February/2021) to receive isotretinoin medication, with any brand names known in Jordan like (ISOSUPRA®, ROACCUTANE®, CURANCE®, RUATINE®,) and met the inclusion criteria were approached and asked to participate in the study. The following are the inclusion criteria:

* Male or female patients aged 18 years or older who were using isotretinoin.
* Patients with a current diagnosis of moderate to severe acne vulgaris.
* Patients who were on or going to receive standard isotretinoin doses (0.5-1mg/kg/day).
* Patients who were willing to participate in the study and to do a follow-up.

Patients with any contraindication to isotretinoin who cannot take the medication and patients who were not willing to participate in the study were excluded as explained in the following:

* Pregnant women and women who intend to become pregnant.
* Breastfeeding women.
* Presence of any renal or hepatic compromise or any pre-existing hyperlipidemia.

The patients were informed about the study objectives, and their voluntary participation, and that withdrawal from the study was possible at any time.

Ethical approval in accordance with regulations was obtained. Institutional Review Board approval was obtained from the IRB at Jordan University of Science and Technology on 27/08/2020. The IRB reference number is (16/134/2020). Patients were asked to sign an informed consent before participating. Participants' privacy was maintained and participants' answers were kept strictly confidential and were never linked to any personal details.

Study Sample and Randomization

The sample size was calculated by OpenEpi, Version 3, open-source calculator-SSCohort/ RCT. The following assumptions were employed: 30% effect size (difference in adherence to recommendation between control (50%) and intervention group (80%)), alpha= 0.05, beta=0.8, and enrollment ratio=1. Accordingly, the minimum sample size of patients needed was 45 patients in each group. In order to adjust for any dropout and to increase the statistical power, the sample size was increased to 200 participants (100 in each group). Enrolled patients were randomized at a ratio of 1:1 using a simple envelope method by flipping a coin.

Data collection

After the informed consent was taken from each patient agreed to participate, the clinical pharmacist measured the level of knowledge about the drug for both groups and measured anxiety and depression score (HADS) at baseline. Then, the participants were randomly assigned to either an intervention group or a control group. Education (recommendations) on isotretinoin was provided by clinical pharmacists to participants in the intervention group only. Both groups received usual routine care (education on isotretinoin provided by a physician). Both patients and the treating physicians were unaware of the assignment to intervention and control groups. Then after three months, a phone call was made to each patient in both groups to measure the extent of knowledge of the drug, the patients' adherence to the drug and the recommendations for appropriate management of side effects, anxiety, and depression score.

Clinical Pharmacist's Role in Study

The first task of the clinical pharmacist was to interview the patients at baseline for both groups to get their responses on the questionnaires of knowledge, and the Hospital Anxiety and Depression Scale (HADS). Second, to educate patients in the intervention group. The education included: the degree of the importance of adherence to the drug and the recommendations, the correct method of taking it, the importance of doing periodic laboratory tests, common side effects, how to properly avoid and deal with side effects, precaution warnings they should pay attention to, and what are the cases in which the drug should be stopped.

Third, the clinical pharmacist distributed brochures in Arabic that contain the most important points about the medication. Finally, after three months, she called all the patients in both groups to get their responses on knowledge about isotretinoin, HADS, and adherence to the medication and recommendations.

Study Questionnaires

The baseline questionnaire was administered in the waiting room of the dermatological clinic, there was no one else present during the interview. The interviewer made sure that the patients understood the questions before answering them. If the patient did not understand a question, the interviewer explained it to him/her. A single interview lasted for approximately 20 - 25 min.

The follow-up questionnaire was administered via phone call. The interviewer confirmed that the patient understood all the questions before answering them. If the patient did not understand a question, the interviewer explained it to him/her. A single interview lasted for approximately 15- 20 min.

Data analysis

After data was collected, the data was entered into Excel worksheets. The responses were coded and entered into SPSS (version 23). Per protocol analysis was used. Descriptive statistics of categorical and continuous variables were calculated. For the categorical variables, the frequency and percentage were calculated, while the arithmetic mean and standard deviation were calculated for continuous variables.

The differences in participants' responses were examined using the Chi-square test (between intervention and control groups) and McNamara's test (between baseline and follow up encounters) for categorical dependent variables as appropriate. For continuous dependent variables, One Way Analysis of Variance (ANOVA) test, independent samples t-test, and Wilcoxon test were performed when applicable. Both Kolmogorov-Smirnov Z and Shapiro-Wilk tests were used to test for normality of continuous variables. The statistical significance level was considered at a p-value ≤ 0.05.

The degree of knowledge and awareness of correct practice was calculated as a total score. McNamara's test was performed to test if there was a significant difference in knowledge before the intervention and after the intervention in the intervention group, and at if there was a significant difference in knowledge between baseline and follow-up in the control group. In addition, independent t-test was used to compare the knowledge score differences (knowledge score at follow up - knowledge score at baseline) between the intervention group and the control group. Linear regression was conducted to evaluate the effect of the educational intervention on the difference in knowledge score adjusting to variables that were unbalanced at baseline.

Patients Adherence to the Recommendations was calculated as a total score for each participant. Average score was evaluated across the intervention and control groups (using t test).

Chi square test was used to compare HADS items at baseline between intervention and control group. Besides, it was used to compare HADS items at follow-up between intervention and control group. Independent t-test was used to compare the HADS score differences (between baseline and at follow up) between the intervention group and the control group.

HADS scores were categorized into three categories based on the abnormality classification; normal (less than eight), borderline abnormal (between eight and eleven) and abnormal (above eleven). Chi square test was used to evaluate the association between HADS score categories and intervention control status at baseline and at follow up.

The percentages (%) of patients' adherence to medication and non-pharmacological adherence were calculated. The reasons behind the patient's non-adherence were themed into three distinct groups (forgetfulness, run out, and unavailability of isotretinoin). The frequency (%) of each group was calculated. Chi-square test was conducted to evaluate the association between adherence status and patient intervention control status.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older who were using isotretinoin.
* Patients with a current diagnosis of moderate to severe acne vulgaris.
* Patients who were on or going to receive standard isotretinoin doses (0.5-1mg/kg/day).
* Patients who were willing to participate in the study and to do a follow-up.

Exclusion Criteria:

* Pregnant women and women who intend to become pregnant.
* Breastfeeding women.
* Presence of any renal or hepatic compromise or any pre-existing hyperlipidemia.
* Patients who were not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Knowledge | 3 months
  The patient knowledge section consisted of ten different questions/items, and each item had two answers (yes/no). Items were coded according to the answer; the correct (adequate) answer was coded as one (1), while the wrong (not adequate) answer was coded as zero (0). So, the knowledge score could take the values of 0 (no knowledge) to 10 (perfect knowledge).
Adherence to the Recommendations | 3 months
  10 items for all patients, and each item had answers (yes/no). Items were coded according to the answer; the correct (adherent) answer was coded as one (1), while the wrong (not adherent) answer was coded as zero (0). The adherence score of patients 'compliance with the recommendations ranged between 0 (least adherent) to 10 (most adherent).

SECONDARY OUTCOMES:
HADS | 3 MONTHS
  consists of fourteen items; seven items each for the depression and anxiety subscale. The score for each item ranges from 0 to 3, and the HADS score ranged from 0 to 21 for depression and the same applied for anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdullah University Hospital, Irbid, Select Region, Jordan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT05839223/Prot_SAP_ICF_000.pdf